CLINICAL TRIAL: NCT07052422
Title: Venetoclax+Decitabine+Busulfan+Fludarabine (VEN+DAC+Bu2Flu4) vs Busulfan+Fludarabine Conditioning Regimen (Bu2Flu5 ) for Older Patients With Myeloid Malignancies Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: VEN+DAC+Bu2Flu4 vs Bu2Flu5 Conditioning Regimen for Elderly Myeloid Malignancies Undergoing Allo-HSCT
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-260
Record Dates: First submitted 2025-06-22; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Older Patients; Myeloid Malignancies; Conditioning; Hematopoietic Stem Cell Transplantation (HSCT)
MeSH Terms: interventions — venetoclax; Decitabine; Busulfan; fludarabine; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VEN+DAC+Bu2Flu4 (Experimental): Venetoclax+Decitabine+Busulfan+Fludarabine
  Interventions: Drug: Venetoclax (VEN); Drug: Decitabine (DAC); Drug: Busulfan (Bu); Drug: Fludarabine (Flu)
- Bu2Flu5 (Active Comparator): Busulfan+Fludarabine
  Interventions: Drug: Busulfan (Bu); Drug: Fludarabine (Flu)

INTERVENTIONS:
Drug: Venetoclax (VEN) — Venetoclax (VEN) was administered at 400mg/day on days -10 to -4.
  Arms: VEN+DAC+Bu2Flu4
Drug: Decitabine (DAC) — Decitabine (DAC) was administered at 20mg/m2/day on days
  -10 to -8.
  Arms: VEN+DAC+Bu2Flu4
Drug: Busulfan (Bu) — Busulfan (Bu) was administered at 3.2 mg/kg/day on days
  -5 to -4.
Drug: Fludarabine (Flu) — Fludarabine (Flu) was administered at 30mg/m2/day on days -5 to -2.
  Arms: VEN+DAC+Bu2Flu4
Drug: Fludarabine (Flu) — Fludarabine (Flu) was administered at 30mg/m2/day on days -6 to -2.
  Arms: Bu2Flu5

SUMMARY:
The purpose of this study is to compare the efficacy and safety of venetoclax+decitabine+busulfan+fludarabine (VEN+DAC+Bu2Flu4) regimen with busulfan+fludarabine (Bu2Flu5) regimen in older patients with myeloid malignancies undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potent curative approach for myeloid malignancies, but outcomes post-transplantation of older population were unsatisfactory. The conditioning regimen is an essential factor affecting outcomes post-transplantation. Currently, the optimal conditioning for older patients with myeloid malignancies remains unclear. Myeloablative conditioning (MAC) regimens like busulfan plus cyclophosphamide, and busulfan plus fludarabine (Bu4Flu4-5) have low relapse rates, but high non-relapse mortality (NRM) is observed in older patients with myeloid malignancies. The development of reduced-intensity conditioning (RIC) regimens such as Bu2Flu5 has decreased NRM and enhanced the feasibility of allo-HSCT in older patients with myeloid malignancies, but it appears to have higher relapse rate. Neither conventional MAC nor RIC regimens benefit older patients with myeloid malignancies. In recent years, some studies reported that the introduction of venetoclax (VEN) or decitabine (DAC) to MAC reduced relapse without increasing NRM in younger patients with high-risk myeloid malignancies. However, whether VEN and DAC combined with RIC regimen reduce relapse without increasing NRM, then improve survival in older patients with myeloid malignancies is unclear. Therefore, we conducted a randomized controlled study to compare the efficacy and safety of VEN+DAC+Bu2Flu4 with Bu2Flu5 in older patients with myeloid malignancies undergoing allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* 60-75 years
* Acute myeloid leukaemia in first complete remission or myelodysplastic syndrome
* Willing to undergo the first allo-HSCT
* Eastern Cooperative Oncology Group performance status of 0-2

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) rate | 2 year
  Will calculate time from random assignment until disease progression or relapse or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) rate | 2 year
  Will calculate time from random assignment until death from any cause.
Relapse incidence | 2 year
  Will calculate time from random assignment until relapse or disease progression.
Non-relapse mortality (NRM) incidence | 2 year
  Defined as death from any cause not subsequent to relapse or disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ling Y, Xuan L, Xu N, Huang F, Fan Z, Guo Z, Xu X, Liu H, Lin R, Yu S, Zhang H, Jin H, Wu M, Liu C, Liang X, Ou R, Zhang Y, Liu X, Qu H, Zhai X, Sun J, Zhao Y, Liu Q. Busulfan Plus Fludarabine Compared With Busulfan Plus Cyclophosphamide for AML Undergoing HLA-Haploidentical Hematopoietic Cell Transplantation: A Multicenter Randomized Phase III Trial. J Clin Oncol. 2023 Oct 10;41(29):4632-4642. doi: 10.1200/JCO.23.00101. Epub 2023 Jun 19. PMID 37335960
- [Background] Rambaldi A, Grassi A, Masciulli A, Boschini C, Mico MC, Busca A, Bruno B, Cavattoni I, Santarone S, Raimondi R, Montanari M, Milone G, Chiusolo P, Pastore D, Guidi S, Patriarca F, Risitano AM, Saporiti G, Pini M, Terruzzi E, Arcese W, Marotta G, Carella AM, Nagler A, Russo D, Corradini P, Alessandrino EP, Torelli GF, Scime R, Mordini N, Oldani E, Marfisi RM, Bacigalupo A, Bosi A. Busulfan plus cyclophosphamide versus busulfan plus fludarabine as a preparative regimen for allogeneic haemopoietic stem-cell transplantation in patients with acute myeloid leukaemia: an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1525-1536. doi: 10.1016/S1470-2045(15)00200-4. Epub 2015 Sep 28. PMID 26429297
- [Background] Devine SM, Owzar K, Blum W, Mulkey F, Stone RM, Hsu JW, Champlin RE, Chen YB, Vij R, Slack J, Soiffer RJ, Larson RA, Shea TC, Hars V, Sibley AB, Giralt S, Carter S, Horowitz MM, Linker C, Alyea EP. Phase II Study of Allogeneic Transplantation for Older Patients With Acute Myeloid Leukemia in First Complete Remission Using a Reduced-Intensity Conditioning Regimen: Results From Cancer and Leukemia Group B 100103 (Alliance for Clinical Trials in Oncology)/Blood and Marrow Transplant Clinical Trial Network 0502. J Clin Oncol. 2015 Dec 10;33(35):4167-75. doi: 10.1200/JCO.2015.62.7273. Epub 2015 Nov 2. PMID 26527780
- [Background] Xuan L, Dai M, Jiang E, Wang Y, Huang F, Fan Z, Xu N, Nie D, Liang X, Chen H, Ye J, Shi P, Liu H, Jin H, Lin R, Yan C, Zhang Y, Sun J, Han M, Liu Q. The effect of granulocyte-colony stimulating factor, decitabine, and busulfan-cyclophosphamide versus busulfan-cyclophosphamide conditioning on relapse in patients with myelodysplastic syndrome or secondary acute myeloid leukaemia evolving from myelodysplastic syndrome undergoing allogeneic haematopoietic stem-cell transplantation: an open-label, multicentre, randomised, phase 3 trial. Lancet Haematol. 2023 Mar;10(3):e178-e190. doi: 10.1016/S2352-3026(22)00375-1. Epub 2023 Jan 23. PMID 36702138
- [Background] Zheng X, Gao H, Lu N, Wang M, Zhang H, Zheng Y, Shen B, Cao Y, Chen X, Zhai W, Wei J, Yang D, Zhang R, Pang A, Feng S, Jiang E, Han M. Efficacy of venetoclax combined with decitabine conditioning regimen for allogeneic hematopoietic stem cell transplantation in high-risk and elderly patients with myeloid neoplasms. Ann Hematol. 2023 Dec;102(12):3603-3611. doi: 10.1007/s00277-023-05500-2. Epub 2023 Oct 25. PMID 37878011